CLINICAL TRIAL: NCT06482281
Title: COVID-19 and Childhood Cancer - Diagnostic Delay, Survival, and COVID-19 Susceptibility
Brief Title: COVID-19 and Childhood Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); The Swedish Childhood Cancer Fund (Unknown)
Responsible Party: Principal Investigator, Giorgio Tettamanti, Senior research specialist, Docent, Karolinska Institutet
Other Study IDs: 2022-06312
Record Dates: First submitted 2024-06-28; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Childhood Cancer; Childhood Leukemia, Acute Lymphoblastic
Keywords: Childhood Cancer; Childhood Cancer Incidence; Childhood Cancer Survival; Childhood Leukemia, Acute Lymphoblastic; Cohort Study; Register Study
MeSH Terms: conditions — COVID-19; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Childhood cancer survivors: Childhood cancer cases (0-19 years old) reported to the national cancer registers from 1971 in Sweden and Denmark, who were alive five years after the cancer diagnosis
- Matched comparisons: Five general population comparisons were randomly selected and matched to the childhood cancer survivors by sex and year of birth
- Siblings: All siblings of the childhood cancer survivors
- Childhood cancer cases: Childhood cancer cases (0-19 years old) reported to the national cancer registers from 2015 in Sweden and Denmark. They will then further divided in three groups: before the pandemic (2015-2019), during the pandemic (2020-2022), and after the pandemic (2022-)

SUMMARY:
The investigators will first examine the impact of the COVID-19 pandemic on childhood cancer patients in Sweden and Denmark, both regarding susceptibility to severe COVID-19 among long-term childhood cancer survivors, and, for those diagnosed with childhood cancer during the pandemic, whether the path through primary care to cancer diagnosis as well as short-term survival has changed. Second, the investigators will study childhood cancer incidence before, during and after the pandemic with the particular aim to test the hypothesis regarding an infectious disease etiology for acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria for studying severe COVID-19 among childhood cancer survivors:

* Childhood cancer cases (age 0-19) diagnosed from 1971 in Sweden and Denmark who were alive five years after diagnosis
* Two different comparisons groups: five age- and sex-matched comparisons for each childhood cancer survivor as well as all siblings of the childhood cancer survivors.
* All childhood cancer survivors, matched comparisons, and siblings of the survivors should be 20+ at the start of 2020.

Inclusion Criteria for studying childhood cancer incidence and survival and number of contacts with healthcare before the childhood cancer diagnosis:

- All children (age 0-19) diagnosed with cancer from 2015 in Sweden and Denmark

Exclusion Criteria:

* No exclusion criteria

Ages: 0 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Childhood cancer cases (age 0-19) diagnosed from 1971 in Sweden and Denmark who were alive five years after diagnosis + their matched comparisons AND all siblings of the childhood cancer survivors
  * All children (age 0-19) diagnosed with cancer from 2015 in Sweden and Denmark
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe COVID-19 | Up to 3 years
  Defined as:
  * death with COVID-19 listed as a cause of death
  * hospitalization, or admission to intensive care unit, because of COVID-19 (main diagnosis) or respiratory problems (main diagnosis) AND COVID-19 as secondary diagnosis
Childhood cancer survival | After three and twelve months after the cancer diagnosis and three years after cancer diagnosis
  Overall survival after a childhood cancer diagnosis
Number of contacts before childhood cancer diagnosis | One year before cancer diagnosis
  Number of healthcare contacts (including primary care) the year before the cancer diagnosis
Childhood cancer incidence | From 2015
  Age standardized incidence rates for childhood cancer and cancer subtypes (particularly acute lymphoblastic leukemia) in Sweden and Denmark during and after the pandemic and compare it to the 5 years preceding the pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Tettamanti, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No